CLINICAL TRIAL: NCT01304355
Title: Kynurenine Pathway Metabolites as Novel Translational Biological Markers of Irritable Bowel Syndrome: Relationship to Gastrointestinal Function, Cognition and Co-morbid Depression
Brief Title: An Assessment of Cognitive Function in Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Collaborators: Science Foundation Ireland (Other); American Neurogastroenterology and Motility Society (Other)
Responsible Party: Professor Ted Dinan, University College Cork
Other Study IDs: APC024-GC/ANMS
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Cognition; Kynurenine Pathway; Gastrointestinal
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma Serum Saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controls: Healthy Control Subjects
- IBS Group: Subjects diagnosed with IBS

SUMMARY:
Irritable bowel syndrome (IBS) is a common disorder affecting up to 20% of the general population. Despite the prevalence of the disorder, it remains poorly understood. This is reflected in a symptom based diagnostic scheme, the lack of a suitable biological marker and inadequate treatment options. Current knowledge suggests the disorder is as a result of a dysregulated brain-gut axis, a complex construct describing the bidirectional communication systems underpinning normal gastrointestinal functioning.

The investigators hypothesize here that the disruption of this brain-gut axis is facilitated by an increased degradation of tryptophan along the kynurenine pathway. This metabolic abnormality has the potential to impact on both GI and CNS signaling through its effects on serotonergic signaling and the impact of metabolites like kynurenic acid and quinolinic acid on cognitive processes respectively.

Previous data from our laboratory indicated increased tryptophan degradation in IBS patients and suggested the metabolites produced as putative biological markers of the condition. In this study the investigators aim to reconcile cognitive impairment in IBS with GI and CNS symptom severity and kynurenine pathway metabolites.

The investigators will establish these baseline measures in IBS compared to control subjects. A battery of cognitive assessments will be carried out using a computerized testing system. Standardized rating scales will be used to assess GI and CNS symptom severity. GC-MS/MS, a recently acquired technology platform in our laboratory, will be used to quantify plasma quinolinic acid levels.

DETAILED DESCRIPTION:
This study is based on the hypothesis that the disruption of this brain-gut axis in irritable bowel syndrome (IBS) is a consequence of increased degradation of tryptophan along the kynurenine pathway. The investigators aim to fully characterize this putative metabolic abnormality and determine its impact on both gastrointestinal (GI) and central nervous system (CNS) signaling by examining the relationship between individual pathway metabolites, GI symptoms and cognitive processing in IBS patients

An increased degradation of tryptophan along the kynurenine pathway has been reported in both depression and IBS (Clarke et al 2009a; Fitzgerald et al 2008; Myint et al 2007). Although such studies have suggested an alteration in the production of quinolinic acid as a consequence of this disruption, actual levels of this NMDA receptor agonist remain to be measured and are essential to the full characterization of pathway disruption. The relevance of this strategy is confirmed by studies that have implicated peripheral quinolinic acid measures as surrogate marker of disease activity in juvenile idiopathic inflammatory myopathies (Rider et al 2002). Moreover it has been demonstrated that increasing plasma levels of this neurotoxic metabolite can influence CNS processes (Yan et al 2005) and that an increased peripheral production of kynurenine can increase central quinolinic acid concentrations (Raison et al 2009a). A correlation between alterations in the kynurenine pathway, GI disturbances and cognitive outcomes remains to be fully defined. In this study, the investigators propose to obtain a complete profile of plasma kynurenine pathway metabolites in IBS patients with and without comorbid depression. Temporal instability in symptom profile is a hallmark of IBS and represents a considerable obstacle to biomarker discovery (Clarke et al 2009b). The preliminary data generated here will potentially be used as the basis for future grant applications that will propose a longitudinal study of these putative biomarker candidates.

BACKGROUND/SIGNIFICANCE

Irritable bowel syndrome (IBS) is a functional gastrointestinal disorder accounting for up to 20% of cases presenting at gastroenterologist clinics in the western world with an unexplained female predominance (Ersryd et al 2007). Although the typical symptoms are commonly experienced in the general population, the abdominal pain and disturbances in defecatory function experienced by IBS sufferers are on a scale that positions the disorder as one of the leading causes of work absenteeism and presenteeism in western societies. Clearly the burden it places on the individual sufferer and society as a whole is substantial and is further compounded by its draining of healthcare resources (Clarke et al 2009b).

Despite the widespread prevalence of the disorder is it still poorly understood and is largely characterized by the lack of a reliable validated biological marker. This is reflected in the reliance on symptom based diagnostic criteria in conjunction with the exclusion of other gastrointestinal disorders (Drossman 2006). Further complications arise in the form of the psychiatric comorbidity so frequently observed among the IBS population (Spiller 2004). It is perhaps unsurprising then that treatment options are inadequate and advances in our understanding of the disorder are urgently required to address the unmet medical needs of its sufferers.

Tryptophan is an essential amino acid and its role as a precursor to many biologically active agents ensures its importance in the consideration of a variety of disease states including schizophrenia (Barry et al 2009; Schwarcz and Pellicciari 2002), depression (Myint et al 2007) and inflammatory bowel disease (Forrest et al 2003). Although much of the attention to date has focused on the production of serotonin from tryptophan, the often-overlooked kynurenine metabolic pathway (Appendix figure 1) consumes over 95% of the available peripheral tryptophan in mammals (Clarke et al 2009a). The first step in this cascade involves the conversion of tryptophan to kynurenine with reports suggesting that the majority of CNS concentrations of the metabolite are drawn from the periphery (Myint et al 2007). This is an important consideration and validates the use of plasma tryptophan metabolites in biomarker studies. This first rate limiting step in the metabolic cascade is catalysed by either the ubiquitous indoleamine-2,3-dioxygenase (IDO) or the largely hepatic based tryptophan 2,3-dioxygenase (TDO). Crucially in the context of stress related disorders like IBS and depression, the activity of both enzymes can be induced by agents which are stress responsive-IDO by inflammatory mediators and TDO by corticosteroids (Ruddick et al 2006).

Once formed, kynurenine essentially participates in two important but alternate metabolic scenarios-one leading to the formation of the neuroprotective kynurenic acid and the other leading to the production of the neurotoxic quinolinic acid (Ruddick et al 2006). The neuroprotective effects of kynurenic acid are attributed to its competitive blockade of the NMDA receptor at the glycine co-agonist site. Conversely quinolinic acid has excititoxic properties due to its potent activation of the NR2A and NR2B NMDA receptor subunits (Schwarcz and Pellicciari 2002). Clearly any imbalance in the production of these bioactive ligands could lead to profound disturbances in CNS glutamatergic signaling and thus affect glutamate-driven behaviours such as learning and memory.

Recent progress in the study of IBS has largely been brought about by a theoretical view of the condition as a disorder of the brain-gut axis (Ohman and Simren 2007). Within this construct, stressful insults are now thought to be integral to the destabilization of normal brain-gut axis signaling. Higher brain centres are involved both in the processing of afferent GI signals and the communication of changes in an individuals emotional state to the gastrointestinal tract (Mayer 2000a; Mayer 2000b). The emotional motor system, consisting of the limbic system and paralimbic structures such as the medial prefrontal cortex, amygdala and hypothalamus, is one such centre. The importance of these structures in the maintenance of normal cognitive function implies that brain-gut axis perturbations could manifest as cognitive impairment across a number of domains.

Other lines of evidence also support an altered neuropsychological state in IBS. An emerging body of research points to the presence of a low grade inflammation in this disorder (Barbara and Stanghellini 2009; Clarke et al 2009b). It has recently been reported that baseline interleukin-6 levels, the cytokine that is most consistently reported to be elevated in IBS (Clarke et al 2009b), is predictive of cognitive symptoms of depression at follow up in a longitudinal study (Gimeno et al 2009). It has also been demonstrated that patients with chronic fatigue syndrome, a disorder that has also been linked with increased inflammatory mediators (Raison et al 2009b), have associated cognitive deficits (Thomas and Smith 2009). Previous studies from our laboratory have highlighted the relationship between the inflammatory profile in IBS and an increased degradation of tryptophan along the kynurenine pathway (Clarke et al 2009a; Fitzgerald et al 2008). Moreover, cancer patients treated by cytokine immunotherapy experience related and persistent cognitive alterations (Capuron et al 2001) and the cognitive alterations accompanying infection are also present in apyretic sick subjects (Capuron et al 1999). The increased tryptophan degradation observed following this immunotherapy is considered to be a key mediator of the resulting neuropsychological alterations (Capuron et al 2002; Raison et al 2009a). Cumulatively, these studies suggest that IBS is a disorder possessing a molecular signature (increased, inflammation and disturbed tryptophan metabolism) indicative of cognitive deficits.

However, despite the uncovering of this molecular signature in IBS, the widespread acceptance of the brain-gut axis model and the high psychiatric comorbidity, a comprehensive cognitive profiling of the IBS patient population has not been performed. The cognitive assessments that have been reported support a cognitive phenotype in the disorder but to date have focused on singular aspects of affective memory performance (Kilkens et al 2005; Kilkens et al 2004) or verbal IQ deficits (Dancey et al 2009). Moreover, there has been, to our knowledge no study correlating cognitive function with mechanistically-oriented biomarkers.

Before the benefits of such a correlation can be accrued however, a more complete assessment of cognitive dysfunction in IBS is urgently required. The Cambridge Neuropsychological Test Automated Battery (CANTAB) is a computerized cognitive assessment program that covers within its remit a broad section of cognitive domains (Fray and Robbins 1996). The battery has been validated in the assessment of cognitive dysfunction across a wide range of disease states including psychiatric disorders such as anxiety (Kaplan et al 2006) and both unipolar and bipolar mood disorders (Elliott et al 1996; Sweeney et al 2000). Insights gained from neuroimaging studies in IBS which highlight the higher brain centres functioning abnormally in the syndrome (Mayer et al., 2008) can be used to inform the initial choice of tests to be applied to IBS subjects. Investigations in other disorders that are reported to have an inflammatory component such as chronic fatigue disorder where assessments of free recall, reaction time and vigilance in conjunction with the Stroop colour-word interference task to measure distraction from irrelevant stimuli have yielded interesting results (Thomas and Smith 2009). The specific executive function assessments which can be applied include the Stocking of Cambridge Task (SOC) which assesses a subject's ability to rearrange a set of balls in a specified minimum number of moves and minimum time and the intradimensional/extradimensional (ID/ED) attentional set shifting task (adapted from the Wisconcin Card Sorting Test (WCST)) used to assess a subjects ability to maintain attention. CANTAB visual memory tasks such as the spatial recognition memory task (SRM) and the paired associates learning task (PAL) can be used to assess deficits in memory (Michopoulos et al 2008). Taken together, these tests are sensitive to dysfunction across a number of different brain regions (Sweeney et al 2000). Recently the cognitive assessments available in the CANTAB battery have been used in conjunction with measures of clinical insight to assess the association between poor insight and cognitive impairment in schizophrenia (Donohoe et al 2009). This may also be relevant to IBS where an increased awareness of and concern about bodily sensations and GI functioning is well established (Posserud et al 2009). It will also be important to rule out alternative explanations for any alterations that are observed included task irrelevant thoughts related to the disease. Few attempts have been made to link such findings to GI symptoms and putative biological marker candidates.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent,
* Be between the ages of 18 and 65 years of age,
* Must be female,
* IBS patients must have a confirmed clinical diagnosis IBS using Rome III criteria
* Healthy subjects must be in generally good health as determined by the investigator
* Pregnant women
* Individuals with known lactose intolerance or immunodeficiency will be excluded

Exclusion Criteria:

* Are less than 18 and greater than 65 years of age,
* Have a significant acute or chronic coexisting illness [cardiovascular, gastrointestinal, immunological, or any condition which contraindicates, in the investigators judgement, entry to the study].
* Having a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include, anti-psychotics and steroids (in healthy and IBS subjects).
* Have evidence of immunodeficiency; bleeding disorder or coagulopathy.
* Subjects may not be receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBS Patients will be recruited from a university database of IBS patients, comprising people who have previously either attended gastroenterology clinics at Cork University Hospital or responded to direct advertisement regarding participation in IBS research.
  Healthy Controls will be recruited from responders to a direct advertisement regarding participation in IBS research
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
CANTAB Assessments | Baseline
  Cognitive assessments using CANTAB, a computerised cognitive assessment package
IBS Symptom Severity | Baseline
  As assessment of IBS symptom severity using validated questionnaires
Kynurenine Pathway Metabolies | Baseline
  Plasma tryptophan, kynurenine, kynurenic acid, quinolinic acid
Glucocorticoids | Baseline
  Plasma/Salivary Cortisol
Cytokines | Baseline
  Plasma Cytokine concentrations
Psychiatric Comorbidity | Baseline
  Psychiatric comorbidity will be assessed according to DSM-IV criteria

SECONDARY OUTCOMES:
Sleep Quality | Baseline
  The potential confounding effect of sleep quality will be established using the Pittsburg Sleep Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Clarke, PhD, Principal Investigator — University College Cork; Timothy G Dinan, Professor, Principal Investigator — University College Cork; John F Cryan, PhD, Principal Investigator — University College Cork
Locations (2):
- Ireland (2):
  - Cork University Hospial, Cork, Cork
  - University College Cork, Cork, Cork

REFERENCES:
- [Background] Barbara G, Stanghellini V. Biomarkers in IBS: when will they replace symptoms for diagnosis and management? Gut. 2009 Dec;58(12):1571-5. doi: 10.1136/gut.2008.169672. No abstract available. PMID 19923339
- [Background] Barry S, Clarke G, Scully P, Dinan TG. Kynurenine pathway in psychosis: evidence of increased tryptophan degradation. J Psychopharmacol. 2009 May;23(3):287-94. doi: 10.1177/0269881108089583. Epub 2008 Jun 18. PMID 18562404
- [Background] Capuron L, Lamarque D, Dantzer R, Goodall G. Attentional and mnemonic deficits associated with infectious disease in humans. Psychol Med. 1999 Mar;29(2):291-7. doi: 10.1017/s0033291798007740. PMID 10218921
- [Background] Capuron L, Ravaud A, Dantzer R. Timing and specificity of the cognitive changes induced by interleukin-2 and interferon-alpha treatments in cancer patients. Psychosom Med. 2001 May-Jun;63(3):376-86. doi: 10.1097/00006842-200105000-00007. PMID 11382265
- [Background] Capuron L, Ravaud A, Neveu PJ, Miller AH, Maes M, Dantzer R. Association between decreased serum tryptophan concentrations and depressive symptoms in cancer patients undergoing cytokine therapy. Mol Psychiatry. 2002;7(5):468-73. doi: 10.1038/sj.mp.4000995. PMID 12082564
- [Background] Clarke G, Fitzgerald P, Cryan JF, Cassidy EM, Quigley EM, Dinan TG. Tryptophan degradation in irritable bowel syndrome: evidence of indoleamine 2,3-dioxygenase activation in a male cohort. BMC Gastroenterol. 2009 Jan 20;9:6. doi: 10.1186/1471-230X-9-6. PMID 19154614
- [Background] Clarke G, Quigley EM, Cryan JF, Dinan TG. Irritable bowel syndrome: towards biomarker identification. Trends Mol Med. 2009 Oct;15(10):478-89. doi: 10.1016/j.molmed.2009.08.001. Epub 2009 Oct 5. PMID 19811951
- [Background] Dancey CP, Attree EA, Stuart G, Wilson C, Sonnet A. Words fail me: the verbal IQ deficit in inflammatory bowel disease and irritable bowel syndrome. Inflamm Bowel Dis. 2009 Jun;15(6):852-7. doi: 10.1002/ibd.20837. PMID 19130620
- [Background] Donohoe G, Hayden J, McGlade N, O'Grada C, Burke T, Barry S, Behan C, Dinan TG, O'Callaghan E, Gill M, Corvin AP. Is "clinical" insight the same as "cognitive" insight in schizophrenia? J Int Neuropsychol Soc. 2009 May;15(3):471-5. doi: 10.1017/S1355617709090559. PMID 19402933
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Elliott R, Sahakian BJ, McKay AP, Herrod JJ, Robbins TW, Paykel ES. Neuropsychological impairments in unipolar depression: the influence of perceived failure on subsequent performance. Psychol Med. 1996 Sep;26(5):975-89. doi: 10.1017/s0033291700035303. PMID 8878330
- [Background] Ersryd A, Posserud I, Abrahamsson H, Simren M. Subtyping the irritable bowel syndrome by predominant bowel habit: Rome II versus Rome III. Aliment Pharmacol Ther. 2007 Sep 15;26(6):953-61. doi: 10.1111/j.1365-2036.2007.03422.x. PMID 17767480
- [Background] Fitzgerald P, Cassidy Eugene M, Clarke G, Scully P, Barry S, Quigley Eamonn MM, Shanahan F, Cryan J, Dinan Timothy G. Tryptophan catabolism in females with irritable bowel syndrome: relationship to interferon-gamma, severity of symptoms and psychiatric co-morbidity. Neurogastroenterol Motil. 2008 Dec;20(12):1291-7. doi: 10.1111/j.1365-2982.2008.01195.x. Epub 2008 Sep 24. PMID 18823288
- [Background] Forrest CM, Gould SR, Darlington LG, Stone TW. Levels of purine, kynurenine and lipid peroxidation products in patients with inflammatory bowel disease. Adv Exp Med Biol. 2003;527:395-400. doi: 10.1007/978-1-4615-0135-0_46. PMID 15206756
- [Background] Fray PJ, Robbins TW. CANTAB battery: proposed utility in neurotoxicology. Neurotoxicol Teratol. 1996 Jul-Aug;18(4):499-504. doi: 10.1016/0892-0362(96)00027-x. PMID 8866544
- [Background] Gimeno D, Kivimaki M, Brunner EJ, Elovainio M, De Vogli R, Steptoe A, Kumari M, Lowe GD, Rumley A, Marmot MG, Ferrie JE. Associations of C-reactive protein and interleukin-6 with cognitive symptoms of depression: 12-year follow-up of the Whitehall II study. Psychol Med. 2009 Mar;39(3):413-23. doi: 10.1017/S0033291708003723. Epub 2008 Jun 4. PMID 18533059
- [Background] Kaplan JS, Erickson K, Luckenbaugh DA, Weiland-Fiedler P, Geraci M, Sahakian BJ, Charney D, Drevets WC, Neumeister A. Differential performance on tasks of affective processing and decision-making in patients with Panic Disorder and Panic Disorder with comorbid Major Depressive Disorder. J Affect Disord. 2006 Oct;95(1-3):165-71. doi: 10.1016/j.jad.2006.04.016. Epub 2006 Jun 21. PMID 16793143
- [Background] Kilkens TO, Honig A, Fekkes D, Brummer RJ. The effects of an acute serotonergic challenge on brain-gut responses in irritable bowel syndrome patients and controls. Aliment Pharmacol Ther. 2005 Nov 1;22(9):865-74. doi: 10.1111/j.1365-2036.2005.02660.x. PMID 16225497
- [Background] Kilkens TO, Honig A, van Nieuwenhoven MA, Riedel WJ, Brummer RJ. Acute tryptophan depletion affects brain-gut responses in irritable bowel syndrome patients and controls. Gut. 2004 Dec;53(12):1794-800. doi: 10.1136/gut.2004.041657. PMID 15542517
- [Background] Mayer EA. Spinal and supraspinal modulation of visceral sensation. Gut. 2000 Dec;47 Suppl 4(Suppl 4):iv69-72; discussion iv76. doi: 10.1136/gut.47.suppl_4.iv69. No abstract available. PMID 11076922
- [Background] Mayer EA, Bradesi S, Chang L, Spiegel BM, Bueller JA, Naliboff BD. Functional GI disorders: from animal models to drug development. Gut. 2008 Mar;57(3):384-404. doi: 10.1136/gut.2006.101675. Epub 2007 Oct 26. PMID 17965064
- [Background] Michopoulos I, Zervas IM, Pantelis C, Tsaltas E, Papakosta VM, Boufidou F, Nikolaou C, Papageorgiou C, Soldatos CR, Lykouras L. Neuropsychological and hypothalamic-pituitary-axis function in female patients with melancholic and non-melancholic depression. Eur Arch Psychiatry Clin Neurosci. 2008 Jun;258(4):217-25. doi: 10.1007/s00406-007-0781-8. PMID 18297425
- [Background] Myint AM, Kim YK, Verkerk R, Scharpe S, Steinbusch H, Leonard B. Kynurenine pathway in major depression: evidence of impaired neuroprotection. J Affect Disord. 2007 Feb;98(1-2):143-51. doi: 10.1016/j.jad.2006.07.013. Epub 2006 Sep 6. PMID 16952400
- [Background] O'Mahony S, Chua AS, Quigley EM, Clarke G, Shanahan F, Keeling PW, Dinan TG. Evidence of an enhanced central 5HT response in irritable bowel syndrome and in the rat maternal separation model. Neurogastroenterol Motil. 2008 Jun;20(6):680-8. doi: 10.1111/j.1365-2982.2007.01065.x. Epub 2008 Jan 13. PMID 18194152
- [Background] O'Mahony SM, Marchesi JR, Scully P, Codling C, Ceolho AM, Quigley EM, Cryan JF, Dinan TG. Early life stress alters behavior, immunity, and microbiota in rats: implications for irritable bowel syndrome and psychiatric illnesses. Biol Psychiatry. 2009 Feb 1;65(3):263-7. doi: 10.1016/j.biopsych.2008.06.026. Epub 2008 Aug 23. PMID 18723164
- [Background] Ohman L, Simren M. New insights into the pathogenesis and pathophysiology of irritable bowel syndrome. Dig Liver Dis. 2007 Mar;39(3):201-15. doi: 10.1016/j.dld.2006.10.014. Epub 2007 Jan 30. PMID 17267314
- [Background] Posserud I, Svedlund J, Wallin J, Simren M. Hypervigilance in irritable bowel syndrome compared with organic gastrointestinal disease. J Psychosom Res. 2009 May;66(5):399-405. doi: 10.1016/j.jpsychores.2008.09.020. Epub 2009 Jan 8. PMID 19379956
- [Background] Raison CL, Dantzer R, Kelley KW, Lawson MA, Woolwine BJ, Vogt G, Spivey JR, Saito K, Miller AH. CSF concentrations of brain tryptophan and kynurenines during immune stimulation with IFN-alpha: relationship to CNS immune responses and depression. Mol Psychiatry. 2010 Apr;15(4):393-403. doi: 10.1038/mp.2009.116. Epub 2009 Nov 17. PMID 19918244
- [Background] Rider LG, Schiffenbauer AS, Zito M, Lim KL, Ahmed A, Zemel LS, Rennebohm RM, Passo MH, Summers RM, Hicks JE, Lachenbruch PA, Heyes MP, Miller FW; Juvenile Dermatomyositis Disease Activity Collaboration Study Group. Neopterin and quinolinic acid are surrogate measures of disease activity in the juvenile idiopathic inflammatory myopathies. Clin Chem. 2002 Oct;48(10):1681-8. PMID 12324484
- [Background] Robbins TW, Arnsten AF. The neuropsychopharmacology of fronto-executive function: monoaminergic modulation. Annu Rev Neurosci. 2009;32:267-87. doi: 10.1146/annurev.neuro.051508.135535. PMID 19555290
- [Background] Ruddick JP, Evans AK, Nutt DJ, Lightman SL, Rook GA, Lowry CA. Tryptophan metabolism in the central nervous system: medical implications. Expert Rev Mol Med. 2006 Aug 31;8(20):1-27. doi: 10.1017/S1462399406000068. PMID 16942634
- [Background] Schwarcz R. The kynurenine pathway of tryptophan degradation as a drug target. Curr Opin Pharmacol. 2004 Feb;4(1):12-7. doi: 10.1016/j.coph.2003.10.006. PMID 15018833
- [Background] Schwarcz R, Pellicciari R. Manipulation of brain kynurenines: glial targets, neuronal effects, and clinical opportunities. J Pharmacol Exp Ther. 2002 Oct;303(1):1-10. doi: 10.1124/jpet.102.034439. PMID 12235226
- [Background] Spiller RC. Irritable bowel syndrome. Br Med Bull. 2005 Mar 14;72:15-29. doi: 10.1093/bmb/ldh039. Print 2004. PMID 15767561
- [Background] Sweeney JA, Kmiec JA, Kupfer DJ. Neuropsychologic impairments in bipolar and unipolar mood disorders on the CANTAB neurocognitive battery. Biol Psychiatry. 2000 Oct 1;48(7):674-84. doi: 10.1016/s0006-3223(00)00910-0. PMID 11032979
- [Background] Thomas M, Smith A. An investigation into the cognitive deficits associated with chronic fatigue syndrome. Open Neurol J. 2009 Feb 27;3:13-23. doi: 10.2174/1874205X00903010013. PMID 19452031
- [Background] Yan E, Castillo-Melendez M, Smythe G, Walker D. Quinolinic acid promotes albumin deposition in Purkinje cell, astrocytic activation and lipid peroxidation in fetal brain. Neuroscience. 2005;134(3):867-75. doi: 10.1016/j.neuroscience.2005.04.056. PMID 16026935